CLINICAL TRIAL: NCT05547984
Title: A Randomized Controlled Trial Comparing Modular Dual Mobility Inserts With Ceramic Multilayer Coating Versus Standard Polyethylene Inserts for Primary Total Hip Arthroplasty (THA) in a Cementless Acetabular Cup
Brief Title: Ceramic Modular Dual Mobility in Primary Total Hip Arthroplasty (THA)
Acronym: CeMoD-prime
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-2203
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Coxarthrosis; Primary
Keywords: Dual Mobility Cup; Total Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Mobility Cup (Experimental): dual mobility articulation
  Interventions: Device: Dual Mobility Cup
- Standard Acetabular component (Active Comparator): standard articulation with polyethylene + vitamin E inlay and metal head
  Interventions: Device: Standard Acetabular component

INTERVENTIONS:
Device: Dual Mobility Cup — Total hip arthroplasty (THA) is a successful and established therapy for coxarthrosis, rheumatic arthritis, hip fractures and femoral head necrosis. The acetabular implant for this arm is the Dual Mobility cup
  Other Names: Total Hip Arthroplasty
  Arms: Dual Mobility Cup
Device: Standard Acetabular component — Total hip arthroplasty (THA) is a successful and established therapy for coxarthrosis, rheumatic arthritis, hip fractures and femoral head necrosis. The acetabular implant for this arm is the standard device with polyethylene + vitamin E inlay and metal head
  Other Names: Total Hip Arthroplasty
  Arms: Standard Acetabular component

SUMMARY:
A randomized controlled trial comparing modular dual mobility inserts with ceramic multilayer coating versus standard polyethylene inserts for primary THA in a cementless acetabular cup

DETAILED DESCRIPTION:
The aim of this study is to show in a randomized controlled trial that cobalt and chromium ion serum levels are comparable to the metal ion levels in patients with standard articulation with metal head. The metal on polyethylene articulation is accepted as standard articulation since many decades, and which is currently in the Czech Republic the most used combination. Most studies which focused on the topic of metal ion release from modular dual mobility systems do not present results of a control group with standard articulation hip implants.

ELIGIBILITY:
Inclusion Criteria:

* Primary coxarthrosis patients indicated for cementless total hip arthroplasty
* Written informed patient consent

Exclusion Criteria:

* Hip trauma or revision surgery
* Rheumatoid or neurologic disease
* BMI >35
* Ongoing oncologic therapy
* Preoperatively elevated Co or Cr serum levels >1.0 µg/L
* Patients with other joint implants, or anticipated need for another joint replacement surgery within the study period
* Acetabular cup size <52 expected
* Patients not able to mentally or physically comply with the study demands and follow-up visits
* Patients <18 years at surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Serum metal ion analysis (Cobalt) | 12 months after surgery
  Cobalt ion levels in blood serum in measured in [µg/L], Comparison between the two groups
Serum metal ion analysis (Chromium) | 12 months after surgery
  Chromium ion levels in blood serum in measured in [µg/L], Comparison between the two groups

SECONDARY OUTCOMES:
Change of functional outcome over three year follow-up period (Harris Hip Score) | 3 months, 12 months and 3 years postoperatively
  The Harris Hip Score (HHS) is one of the most used scores in total hip arthroplasty, mainly combining range of motion questions with questions regarding daily life activities. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100, any result <70 is considered a poor result; The HHS is an outcome measure administered by a qualified health care professional, such as a physician or a physical therapist.
Gait analysis over time | preoperative, 3 months and 12 months postoperatively
  The gait lab analysis involves a high amount of recorded data and variables. Gait lab analyses are performed with the patients between the preoperative state, 3 months after surgery and 1 year postoperative. The Gait Profile Score (GPS) is used as a measure for the deviation in gait kinematics from a healthy patient population to compare the two treatment groups.
  Lower score values can be considered as a sign of better restoration of the physiological gait kinematics.
Development of Patient satisfaction with surgery result over time | at three examinations during Follow-Up (3 months postop, 1 year postop, 3 years postop)
  Patient is asked for satisfaction with surgery result with a 4-point scale: very satisfied, satisfied, unsatisfied, very unsatisfied
Radiologic Evaluation: Cup Inclination over time | immediately postoperative, 3 months, 12 months and 3 years postoperative
  Inclination is the orientation of the cup in the coronal plane. The target acetabular cup inclination is a "safe zone" between 30-50° abduction (assessed on antero-posterior (ap) x-rays of the hip). The comparison of the intraoperatively achieved inclination and the inclination at different follow-up examinations allows prediction on longterm success.
Radiologic Evaluation: center of rotation | immediately postoperative, 3 months, 12 months and 3 years postoperative
  Centre of Rotation (CoR) is defined as the zero position for the measurement of potential cup migration. Horizontal: Distance of CoR to ipsilateral teardrop; Vertical: Distance CoR to Inter-teardrop line; The comparison of the intraoperatively center of rotation and the center of rotation at different follow-up examinations allows prediction on longterm success.
Radiologic Evaluation: Radiolucencies around the cup | over follow-up period 3 months, 12 months and 3 years postoperative
  Bony Osseointegration or conspicuous features of the cup are assessed on anterior-posterior and lateral x-rays of the cup and will be analysed according to the zones defined by Charnley. "Charnley" zones of the acetabular component are distinct zones used in assessment of aseptic loosening in total hip joint replacements. The radiolucencies are categorized to "none", "less than or equal to 2mm" and "more than 2 mm"
Radiological Outcome: Heterotopic Ossification | over follow-up period 3 months, 12 months and 3 years postoperative
  Brooker classification divides heterotopic ossifications that form following total hip replacement to four classes. Class I: islands of bone within soft tissues around hip; Class II: bone spurs in pelvis or proximal end of femur leaving ≥1 cm between the opposing bone surfaces; Class III: bone spurs that extend from pelvis or the proximal end of femur, which reduce the space between the opposing bone surfaces to <1cm; Class IV: ankylosis of the hip on x-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Masaryk Hospital, Ústí nad Labem, Czechia